CLINICAL TRIAL: NCT01863680
Title: Open-label, Single-arm, Multicenter Phase III Trial to Evaluate the Efficacy and Safety of COL-1620 8% Vaginal Progesterone Gel for Luteal Phase Support in In-vitro Fertilization and Embryo Transfer (IVF/ET) Cycles in Japanese Women
Brief Title: Phase 3 Trial to Evaluate the Efficacy and Safety of COL-1620 Vaginal Progesterone Gel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR200113_001
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Luteal Hormone Supplementation in In-vitro Fertilization; Embryo Transfer
Keywords: Infertility; COL-1620; progesterone gel; Fertilization in Vitro; Embryo Transfer
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone; Follicle Stimulating Hormone; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COL-1620 (Experimental)
  Interventions: Drug: COL-1620; Drug: Gonadotropin-releasing hormone (GnRH) analogue; Drug: Follicle-stimulating hormone (FSH); Drug: Human Chorionic Gonadotropin (hCG)

INTERVENTIONS:
Drug: COL-1620 — The subjects will be administered with COL-1620 vaginal progesterone gel (1.125 grams of progesterone gel containing 90 milligram that is 8 percent [%] gel) vaginally once daily, from the day of ovum pick-up (OPU) until Week 12.
Drug: Gonadotropin-releasing hormone (GnRH) analogue — Subjects will undergo conventional controlled ovarian stimulation (COS) therapy for in-vitro Fertilization and Embryo Transfer (IVF/ET) according to the Investigator's discretion using GnRH analogue (agonist or antagonist) preparation.
Drug: Follicle-stimulating hormone (FSH) — Subjects will undergo conventional COS therapy for IVF/ET according to the Investigator's discretion using FSH containing preparation.
Drug: Human Chorionic Gonadotropin (hCG) — Subjects will undergo conventional COS therapy for IVF/ET according to the Investigator's discretion using hCG preparation.

SUMMARY:
The primary objective of this trial is to demonstrate the non-inferiority of the clinical pregnancy rate per embryo transfer to the historical standard value in in-vitro fertilization (IVF)/embryo transfer (ET) cycles in Japan (Japan Society of Obstetrics and Gynecology [JSOG] 2009 registry data: 24.3 percent [%]). The secondary objectives of this trial are to assess the biochemical pregnancy rate per ET, pharmacokinetics, and safety of COL-1620.

ELIGIBILITY:
Inclusion Criteria:

* Japanese race
* Woman with a history of infertility and in whom In-vitro fertilization and embryo transfer (IVF/ET) is indicated
* The controlled ovarian stimulation (COS) therapy is gonadotropin-releasing hormone (GnRH) analogue (agonist or antagonist) in combination with a follicle-stimulating hormone (FSH) containing preparation
* Healthy premenopausal woman aged between 20 and 45 years (inclusive) and wishing to conceive
* Body mass index (BMI) of 17.0 to 25.0 kilogram per square meter (kg/m^2) (inclusive)
* A negative pregnancy test (urinary beta-human chorionic gonadotropin [hCG]) prior to starting COS
* Normal cervical smear result (Papanicolaou [PAP] test: Negative for Intraepithelial Lesion or Malignancy [NILM] or [Atypical Squamous Cells of Undetermined Significance {ASC-US} and Human Papillomavirus {HPV} negative]) within 12 months prior to the date of informed consent. If not available, a cervical smear and HPV test will be performed as part of Screening
* No clinically significant abnormal findings in the screening hematology, biochemistry and urinalysis parameters
* Full comprehension of the study and voluntary written informed consent obtained in writing prior to any trial-related activities

Exclusion Criteria:

* History of recurrent pregnancy loss (defined as 3 or more previous spontaneous abortions)
* History of 3 or more consecutive cancelled or failed (no clinical pregnancy) IVF/ET cycles
* Abnormal hemorrhage of the reproductive tract of undetermined origin
* Any contraindication to being pregnant and/or carrying a pregnancy to term (for example, malformations of sexual organs or fibroid tumors of the uterus incompatible with pregnancy)
* Uterine myoma requiring treatment
* Extra-uterine pregnancy within the last 3 months prior to the date of informed consent
* History or presence of intracranial tumor (for example, hypothalamic or pituitary tumor)
* Presence of or suspected gonadotropin- or estrogen-dependent malignancy (for example, ovarian, uterine or mammary carcinoma)
* Ovarian enlargement or cyst of unknown etiology
* Breast-feeding or lactation
* History of severe Ovarian Hyperstimulation Syndrome (OHSS) (Classification of OHSS Severity, as per Japan Reproductive/Endocrine Working Group)
* Known Human Immunodeficiency Virus (HIV)-positive status, or a history of or current active infection with Hepatitis B or C
* Known allergy or hypersensitivity to progesterone preparations or gonadotropin preparations and/or their excipients, or any contraindication to receive medication for controlled ovarian stimulation (for example, gonadotropin, GnRH analogues, combined oral contraceptive pill, as appropriate)
* History of or suspected alcohol or substance abuse within 5 years prior to the date of informed consent
* Clinically significant systemic disease (for example, insulin-dependent diabetes, epilepsy, severe migraine, acute porphyria, hepatic, renal or cardiovascular disease, severe corticosteroid-dependent asthma)
* Active thrombophlebitis, thromboembolic disorder or cerebral apoplexy, or a history of such conditions
* Other significant disease that in the Investigator's or Sub-Investigator's opinion would exclude the subject from the trial
* Participation in another clinical trial within 3 months prior to the date of informed consent or simultaneous participation in another clinical trial
* Legal incapacity or limited legal capacity

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., Japan
Locations (5):
- Japan (5):
  - Research site, Fujimino
  - Research site, Kobe
  - Research site, Osaka
  - Research site, Sagamihara
  - Research site, Yokohama, Kanagawa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject/Last subject (signed informed consent form [ICF]): 22 Jul 2013/02 Jun 2014; Study completed: 14 Oct 2014; Data base lock: 12 Nov 2014.
Pre-assignment Details: A total of 195 subjects were screened and 178 subjects were enrolled in the trial; 169 subjects started controlled ovarian stimulation (COS) treatment and 149 subjects received at least 1 dose of investigational medicinal product (IMP), 123 subjects have undergone in-vitro fertilization/ embryo transfer (IVF/ET).
Groups:
- COL-1620: The subjects were administered with COL-1620 vaginal progesterone gel (1.125 grams of progesterone gel containing 90 milligram that is 8% gel) vaginally once daily, from the day of ovum pick-up (OPU) until Week 12 or until the confirmation of miscarriage or extra-uterine pregnancy, or a negative pregnancy test whichever was earlier.
  Subjects had undergone conventional controlled ovarian stimulation (COS) therapy for in-vitro Fertilization and Embryo Transfer (IVF/ET) according to the Investigator's discretion using Gonadotropin-releasing hormone (GnRH) analogue (agonist or antagonist) preparation, follicle-stimulating hormone (FSH) or human chorionic gonadotropin (hCG).
Period: Overall Study
Arm/Group | COL-1620
Started | 178
Subjects Started COS Treatment | 169
Subjects Received hCG Injection | 162
Subjects Received Study Drug | 149
Subjects Who Have Undergone IVF/ET | 123
Completed | 121
Not Completed | 57
Not completed — Adverse Event | 17
Not completed — Risk of OHSS | 17
Not completed — Spontaneous pregnancy | 2
Not completed — Withdrawal by Subject | 1
Not completed — Did not undergo IVF/ET | 14
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all the subjects who received at least one dose of study drug.
Groups:
- COL-1620: The subjects were administered with COL-1620 vaginal progesterone gel (1.125 grams of progesterone gel containing 90 milligram that is 8% gel) vaginally once daily, from the day of ovum pick-up (OPU) until Week 12 or until the confirmation of miscarriage or extra-uterine pregnancy, or a negative pregnancy test whichever was earlier.
  Subjects had undergone conventional controlled ovarian stimulation (COS) therapy for in-vitro fertilization and embryo transfer (IVF/ET) according to the Investigator's discretion using GnRH analogue (agonist or antagonist) preparation, follicle-stimulating hormone (FSH) or human chorionic gonadotropin (hCG).
Arm/Group | COL-1620
Number analyzed (Participants) | 149
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.41 (3.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pregnancy Rate Per Embryo Transfer
Description: Clinical pregnancy was defined as the presence of a fetal sac on transvaginal ultrasound (TVUS) during Week 5 or the presence of an extra-uterine pregnancy (as confirmed during surgery or by 2 positive serum beta-human chorionic gonadotropin (beta-hCG) results from Week 5). The clinical pregnancy rate was calculated as number of subjects who were clinically pregnant divided by the number of subjects who had at least 1 embryo transferred.
Time Frame: Week 5 post embryo transfer (2-6 days after Ovum Pick-up [OPU])
Population: The intention-to-treat subjects included all the subjects who underwent IVF/ET.
Measure: Number; unit: Percentage of pregnancy/embryo transfer
Arm/Group | COL-1620
Number analyzed (Participants) | 123
Percentage of pregnancy/embryo transfer | 28.5

2. Secondary Outcome: Biochemical Pregnancy Rate Per Embryo Transfer
Description: Biochemical pregnancy was defined as any miscarriage without any evidence of a fetal sac on TVUS during Visit 6 (Week 5), but with a positive serum beta-hCG pregnancy test result at Visit 5 (Day 14+/-3). Biochemical pregnancy rate was calculated as the number of subjects who had no fetal sac observed during Visit 6 (Week 5) TVUS assessment or subjects who had a positive serum pregnancy test at Visit 5 (Day 14+/-3) and no data recorded at Visit 6 (Week 5) divided by the number of subjects who has at least 1 embryo transferred.
Time Frame: Week 5 post embryo transfer (2-6 days after Ovum Pick-up [OPU])
Population: The intention-to-treat subjects included all the subjects who underwent IVF/ET.
Measure: Number; unit: Percentage of pregnancy/embryo transfer
Arm/Group | COL-1620
Number analyzed (Participants) | 123
Percentage of pregnancy/embryo transfer | 7.3

3. Secondary Outcome: Serum Progesterone Level
Description: Two pharmacokinetic (PK) samples were collected per subject for the measurement of serum progesterone concentrations; 1st sample at Visit 2-2 (prior to hCG administration) and second sample during Visit 5 (Day 14+/-3, 7 hours after the morning of investigational medicinal product administration).
Time Frame: Visit 2-2 (Prior to hCG administration) and Visit 5 (Day 14+/-3)
Population: The PK analysis set included all subjects who had serum beta-hCG pregnancy test performed at Visit 5 (Day 14+/-3), who had two progesterone concentrations at Visit 2-2 and Visit 5, and who had no relevant problems for compliance of administration until Visit 5. "n" signifies the number of subjects who were evaluable in each category, respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | COL-1620
Number analyzed (Participants) | 121
nanogram per milliliter (ng/mL)
  Subjects with +ve serum beta-hCG: Visit 2-2 (n=44) | 1.023 (0.414)
  Subjects with +ve serum beta-hCG: Visit 5 (n=44) | 61.508 (76.206)
  Subjects with -ve serum beta-hCG: Visit 2-2 (n=77) | 0.988 (0.471)
  Subjects with -ve serum beta-hCG: Visit 5 (n=77) | 7.765 (3.202)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration up to Week 15
Description: Safety analysis population included all the subjects who received at least one dose of study drug.
Arm/Group | COL-1620
Serious Adverse Events (participants affected / at risk) | 5/149
Other Adverse Events (participants affected / at risk) | 92/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COL-1620 (N=149)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COL-1620 (N=149)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Asthenopia (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain lower (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 2
Anal fissure (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 10
Faeces soft (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Cystitis (Infections and infestations) | 1
Escherichia vaginitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Genital candidiasis (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 8
Vulvitis (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 7
Arthropod sting (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Foreign body (Injury, poisoning and procedural complications) | 2
Injury corneal (Injury, poisoning and procedural complications) | 1
Urine ketone body present (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness postural (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Migraine (Nervous system disorders) | 1
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 3
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 9
Pregnancy of unknown location (Pregnancy, puerperium and perinatal conditions) | 1
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Cervical polyp (Reproductive system and breast disorders) | 2
Genital haemorrhage (Reproductive system and breast disorders) | 3
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1
Hyperreactio luteinalis (Reproductive system and breast disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 6
Ovarian enlargement ' (Reproductive system and breast disorders) | 2
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 29
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
This study was not a randomized controlled study and did not included an active control arm, however it was designed to allow for comparison with historical IVF-ET data from Japan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study as a whole will be published prior to any individual investigator publications. It is required that copies of all papers, abstracts, articles, etc. that contain study data are to be forward to the Sponsor for review 30 days prior to submission for publication.